CLINICAL TRIAL: NCT06537076
Title: A Randomized, Double-blind, Phase IIa Clinical Trial to Study the Safety and Efficacy of AR1005 in Patients with Lewy Body Disease
Brief Title: Safety and Efficacy of AR1005 in Patients with Lewy Body Disease
Acronym: AR1005
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Samjin Pharmaceutical Co., Ltd. (Industry); AriBio Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Byoung Seok Ye, Associate Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR1005-KRP2-01
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Lewy Body Dementia
Keywords: Lewy body dementia; DLB
MeSH Terms: conditions — Lewy Body Disease | interventions — Appointments and Schedules; Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): AR1005 50 mg BID will be administered with rivastigmine 3 mg BID for 20 weeks.
  Interventions: Drug: AR1005; Drug: Rivastigmine 3 mg
- Placebo (Placebo Comparator): Placebo BID will be administered with rivastigmine 3 mg BID for 20 weeks.
  Interventions: Drug: Placebo; Drug: Rivastigmine 3 mg

INTERVENTIONS:
Drug: AR1005 — AR1005 inhibits sodium currents by selective binding to the inactive sodium channel, suppressing the release of the excitatory amino acid, glutamate.
  Other Names: Scheduled for future release
  Arms: Experimental
Drug: Placebo — Matching placebo for AR1005 to be administered BID for 20 weeks
  Arms: Placebo
Drug: Rivastigmine 3 mg — 3mg Rivastigmine will be administered BID for both active and placebo groups

SUMMARY:
This study is a phase 2a, single-center, double-blind and randomized clinical trial that evaluates the safety and efficacy of AR1005 administration in 60 patients with cognitive impairment due to Lewy body disease. The study evaluates whether the administration of AR1005 in patients with cognitive impairment due to Lewy body disease has the effect of improving cognitive function, behavioral psychological symptoms, cognitive fluctuations, movement, brain waves and brain activity.

DETAILED DESCRIPTION:
60 patients will be randomized into either active or placebo groups (1:1). Both groups will concurrently receive standard treatment with rivastigmine for 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* men and women over the age of 60

  * Communication in Korean is possible and the purpose and process of the study are fully understood and agreed

    * Total score of 26 points or less in the simplified mental health assessment (K-MMSE)

      * Dementia Clinical Evaluation Scale (CDR) Total score of 0.5 or higher

        * Medical history, neurological examination, hematologic examination, Seoul neuropsychological examination 2nd edition, brain magnetic resonance imaging suspected of cognitive impairment due to dementia with Lewy bodies as the cause of cognitive decline

          i. Lewy body dementia
          1. In accordance with the guidelines for the 4th report of the Dementia with Lewy Bodies Consortium (DLBC) published in 2017, if it falls under Probable Dementia with Lewy Bodies
          2. Required Requirements

             1. Dementia, defined as cognitive decline that progresses sufficiently to impair normal social and professional functions or daily life
             2. Defects in attention, enforcement, and space-time capabilities are noticeable in the inspection
          3. Core clinical features

             1. variation in cognitive function
             2. vision
             3. Parkinson's syndrome: One or more manifestations of sinusitis, stable progress, or stiffness
             4. REM sleep behavior disorder
          4. Indicative biomarker

             1. Decreased intake of dopamine carrier PET-phase nuclear
             2. [I-123]-MIBG myocardial scintigraphy intake decreased
             3. REM sleep behavior disorder according to polymorphic test
          5. In the case of two or more key aspects, or one or more key clinical features and one or more indicative biomarkers are satisfied

             ii. Bulb Lewy body dementia (Prodromal DLB)

          <!-- -->

          1. If it falls under the Probable MCI-LB with a mild cognitive impairment according to the criteria for diagnosing precursor Lewy body dementia announced in 2020
          2. Required Requirements

             a. cognitive decline observed when judged by the patient, guardian, or clinician b. Objective cognitive decline (although it is not related to any cognitive domain, it should be mainly related to the deterioration of execution function and space-time ability)
          3. Core clinical features

             1. variation in cognitive function
             2. vision (nap, dazed, same document, angry)
             3. Parkinson's syndrome: One or more manifestations of sinusitis, stable progress, or stiffness
             4. REM sleep behavior disorder
          4. Indicative biomarker

             a. Decreased intake of dopamine carrier PET-phase nuclear b. [I-123]-MIBG myocardial scintigraphy intake decreased c. REM sleep behavior disorder according to polymorphic test
          5. The leading mild cognitive impairment due to dementia with Lewy bodies has two or more key features or satisfies one or more key clinical features and one or more indicative biomarkers

             ⑥ Patients with caregivers who are in regular contact with the subject (Note: caregivers may support the subject during the clinical trial [compliance supervision and reporting of the subject's status], defined as those who spend at least 8 hours per week with the subject)

             ⑦ Patients who can walk or move with walking aids (i.e., walkers, canes, or wheelchairs)

             ⑧ Patients with sufficient vision, hearing, language skills, motor skills, and comprehension to follow the examination procedure as judged by the tester (Aids such as glasses and hearing aids are allowed)

             ⑨ an examination Patients who have voluntarily decided to participate in this clinical trial and obtained the consent of the subject in writing from both the subject and the subject's legal representative (where written consent is not available, the tester shall keep a record of the matters that the subject has verbally agreed to participate in the trial)

             Exclusion Criteria:
* In hematologic and brain magnetic resonance imaging tests conducted within 6 months, other causes of cognitive decline such as neurosyphilis, hypo/hyper-throidism, metabolic encephalopathy, brain tumor, acute cerebral hemorrhage, acute cerebral infraction, and Wernicke's encephalopathy are suspected

  * Subjects who are or are suspected of having an irritable allergy to AR1005-KRP2-01

    * If you are already on antistatic medication

      * A person who cannot perform a brain magnetic resonance image (but if there is a brain magnetic resonance image taken within one year, the brain magnetic resonance image can be omitted)

        * voluntary Employees directly involved in this clinical study or their immediate family members who find it difficult to participate

          * If there is a history of psychiatric disorders: major effective disorder, schizophrenia, schizo-effective disorder

            ⑦ If an electroencephalogram cannot be performed

            ⑧ Patients who are already taking acetylcholinesterase inhibitor (donepezil and rivastigmine) or taking it in patch form (but can change to rivastigmine PO to participate in the study)

            ⑨ Patients with moderate to severe liver disorder (Child-Pugh grade B) and dialysis due to decreased renal functiona patient with end-stage renal impairment receiving

            ⑩ Patients discontinued administration due to aseptic meningitis associated with AR1005-KRP2-01

            ⑪ Patients with genetic problems such as galactose intolerance, lactose-degrading enzyme deficiency, or glucose-galactose absorption disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Dementia Rating-Sum Of Boxes (CDR-SOB) at Week 20 | 20 Weeks
  The CDR-SOB score ranges from 0 to 18, with 0 indicating no dementia symptoms and 18 indicating severe dementia. Higher scores on the CDR-SOB reflect a worse outcome, as they indicate more severe dementia symptoms.

SECONDARY OUTCOMES:
Change in K-MMSE over 20 weeks | 20 Weeks
  Change in Korean-Mini Mental State Examination (K-MMSE) over 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Byoung Seok Ye, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: Will be made available after the study is completed.
Access Criteria: Access will be provided to qualified researchers affiliated with recognized institutions, who have a valid research plan and appropriate ethical approvals.